CLINICAL TRIAL: NCT05977075
Title: Training "Unstuck and On Target! Second Edition" Versus Training "ApisMela"
Brief Title: Group Intervention on Executive Function in Children With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Fondazione di Comunità di Messina onlus (Unknown)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CNR-IRIB-PRO-2023-003
Record Dates: First submitted 2023-07-14; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: autism; children; executive functions
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "ApisMela/Unstuck" Group (Experimental): Six children belonging to the experimental group. ApisMela training teaches to focus on the purpose of the task, check that you understand it, and make explicit the procedures to be implemented. Being a crossover clinical trial, the group ending with the ApisMela protocol continues with the Ustuck protocol.
  Interventions: Other: ApisMela protocol; Other: "Unstuck and on Target" protocol
- "Unstuck/ApisMela" Group (Experimental): Six children belonging to the experimental group. Unstuck protocol teaches people to be more flexible, skillful in planning and goal-oriented. Being a crossover clinical trial, the group ending with the Unstuck protocol continues with the ApisMela protocol.
  Interventions: Other: ApisMela protocol; Other: "Unstuck and on Target" protocol

INTERVENTIONS:
Other: ApisMela protocol — The activities and games proposed by this protocol are offered in a sequence characterized by increasing complexity. The same function is stimulated with varied tasks because the repetitiveness of the same task negatively affects skill generalization. ApisMela training teaches to focus on the purpose of the task, check that you understand it, and make explicit the procedures to be implemented. Language plays a crucial role, participants are encouraged to use speech as a tool for attention regulation and cognitive processing. It's divided into 20 sessions: a weekly group meeting of one hour and thirty.
Other: "Unstuck and on Target" protocol — The protocol teaches people to be more flexible, skillful in planning and goal-oriented. It is useful for moving more easily from one topic to another and from one task to another, considering new ideas or another person's point of view, generalizing skills learned across contexts so that teachers, parents and therapists can focus more on educational aspects and less on behavioral management. It is divided into 20 sessions: a weekly group meeting of one hour and thirty minutes. A homework sheet is provided for each session to consolidate the skill learned and generalize it outside the work setting. Parents have an active role in performing the task.

SUMMARY:
Autism is a developmental disorder characterized by difficulties in social communication, repetitive behaviors, and social interaction. A key aspect of autism concerns executive functions, which are a set of cognitive processes that regulate attention, planning, inhibition, and impulse control. These functions are often impaired in children with autism, affecting their learning and daily functioning.

The present protocol aims to test the first absolute and then comparative effectiveness of two executive function development programs: the "APISMELA" training and the "UNSTUCK & ON TARGET! SECOND EDITION". Two groups will be held at the same time and will conduct the two programs in reverse order. In fact, the protocol is divided into two phases.

Participants subjected to the APISMELA group, finished the intervention sessions will conduct an interim evaluation and then begin the intervention phases of the UNSTUCK & ON TARGET! SECOND EDITION protocol.

Participants subjected to the UNSTUCK & ON TARGET! SECOND EDITION group, finished the intervention sessions will conduct an interim evaluation and then begin the intervention phases of the APISMELA protocol.

Group intervention programs were chosen for two reasons: group intervention compared with individual intervention have lower costs for patients and their families and thus higher overall social acceptability. The second is that group intervention within the social-constructivist paradigm, to which the two chosen programs belong, becomes a fundamental resource for stimulating that augmentative learning that is a source of development on the cognitive and conceptual levels for human beings.

ELIGIBILITY:
Inclusion Criteria:

* Children with diagnosis of autism and autism spectrum disorder

Exclusion Criteria:

* Presence of other medical disorders

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Wechsler Intelligence Scale for Children Fourth edition (WISC-IV) | The evaluation session will be scheduled pre-intervention (T0). The test needs approximately 65-80 minutes to complete.
  Wechsler Intelligence Scale for Children Fourth edition (WISC-IV) is a clinical tool for assessing the cognitive abilities of children and young people between the ages of 6 years and 16 years and 11 months.
  The WISC-IV scales are as follows:
  index of verbal comprehension (ICV), range weighted scores (min 46 - max154); index visuoperceptual reasoning (IRP), range weighted scores (min 41- max 159); index working memory (IML) range weighted scores (min 46 - max 154); processing speed index (IVE) range weighted scores (min 47 - max 153); intelligence quotient IQ (min 40 - max 160). For each sub-scale higher score corresponds to better performance.
Changes in NEuroPSYcology second edition (NEPSY-II) evaluations | The tests will be scheduled pre intervention (T0), at 6 months (T1) and at the study conclusion,about 1 year (T2).The T1 and T2 evaluations were conducted to determine whether the protocols carried out made a change.The test needs about 120-180 minutes.
  NEuroPSYcology second edition (NEPSY-II) is the most internationally known battery for assessing neuropsychological development in developmental age.
  Each NEPSY-II test provides raw scores that must be converted into scalar scores (min 1 - max 19) or percentile scores (min <2% - max >75%) according to the conversion tables in the manual. For each sub-scale higher scores correspond to better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nydén, A., Gillberg, C., Hjelmquist, E., & Heiman, M. (1999). Executive function/attention deficits in boys with Asperger syndrome, attention disorder and reading/writing disorder. Autism, 3(3), 213-228.
- [Background] Jolles DD, Crone EA. Training the developing brain: a neurocognitive perspective. Front Hum Neurosci. 2012 Apr 9;6:76. doi: 10.3389/fnhum.2012.00076. eCollection 2012. PMID 22509161
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, 5th ed.; American Psychiatric Publishing: Washington, DC, USA, 2013.
- [Background] Wilson TD, Reinhard DA, Westgate EC, Gilbert DT, Ellerbeck N, Hahn C, Brown CL, Shaked A. Social psychology. Just think: the challenges of the disengaged mind. Science. 2014 Jul 4;345(6192):75-7. doi: 10.1126/science.1250830. PMID 24994650
- [Background] Kenworthy L, Anthony LG, Naiman DQ, Cannon L, Wills MC, Luong-Tran C, Werner MA, Alexander KC, Strang J, Bal E, Sokoloff JL, Wallace GL. Randomized controlled effectiveness trial of executive function intervention for children on the autism spectrum. J Child Psychol Psychiatry. 2014 Apr;55(4):374-83. doi: 10.1111/jcpp.12161. Epub 2013 Nov 21. PMID 24256459
- [Background] Orsolini, Margherita & Melogno, Sergio & Santese, Angela & Toma, Chiara & Latini, Nausica & Salomone, Samantha & Andreagiovanni, Jacopo. (2019). "Pensando si Impara" STIMOLARE L'ATTENZIONE, LE FUNZIONI ESECUTIVE E LA MEMORIA DI LAVORO NEI BAMBINI CON BISOGNI EDUCATIVI SPECIALI.
- [Background] Dickson KS, Aarons GA, Anthony LG, Kenworthy L, Crandal BR, Williams K, Brookman-Frazee L. Adaption and pilot implementation of an autism executive functioning intervention in children's mental health services: a mixed-methods study protocol. Pilot Feasibility Stud. 2020 Apr 27;6:55. doi: 10.1186/s40814-020-00593-2. eCollection 2020. PMID 32699642
- [Background] Cannon J, O'Brien AM, Bungert L, Sinha P. Prediction in Autism Spectrum Disorder: A Systematic Review of Empirical Evidence. Autism Res. 2021 Apr;14(4):604-630. doi: 10.1002/aur.2482. Epub 2021 Feb 11. PMID 33570249